CLINICAL TRIAL: NCT00743535
Title: A Comparison in Terms of Efficacy and Safety Between Transobturator and Transvaginal Tape Performed at the Same Time of Anterior Defect Correction With Mesh
Brief Title: Anterior Defect Correction With Mesh Plus Treatment of Stress Incontinence With Transobturator or Transvaginal Approach
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment rate.
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Stefano Palomba, Associate Professor, University Magna Graecia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03/2008
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Cystocele; Stress Urinary Incontinence
Keywords: Cystocele; Mesh; Prolapse; Sling; Stress incontinence; Surgery; TOT; TVT; Treatment
MeSH Terms: conditions — Cystocele; Urinary Incontinence, Stress; Prolapse

ARMS (2):
- 1 (Experimental): Transobturatory correction of anterior defect plus TOT
  Interventions: Procedure: Transobturatory correction of anterior defect plus TOT
- 2 (Active Comparator): Longitudinal vaginal incision 1 cm far from esternal urethral meatus. Bladder dissecting and identification of ischiatic spines. Bilateral transobturator insertion of anterior mesh through high and low trans-obturatory approach. Mesh anchorage.
  Small incision sites at sovrapubic level. Bilateral retropubic insertion of mesh by means of mono-use needle.
  Interventions: Procedure: Transobturatory correction of anterior defect plus TVT

INTERVENTIONS:
Procedure: Transobturatory correction of anterior defect plus TOT — Longitudinal vaginal incision 1 cm far from esternal urethral meatus. Bladder dissecting and identification of ischiatic spines. Bilateral transobturator insertion of anterior mesh through high and low trans-obturatory approach. Mesh anchorage.
  Small incision sites in the femoral/pelvic fold. Bilateral transobturator insertion of mesh by means of mono-use needle
  Arms: 1
Procedure: Transobturatory correction of anterior defect plus TVT — Longitudinal vaginal incision 1 cm far from esternal urethral meatus. Bladder dissecting and identification of ischiatic spines. Bilateral transobturator insertion of anterior mesh through high and low trans-obturatory approach. Mesh anchorage.
  Small incision sites at sovrapubic level. Bilateral retropubic insertion of mesh by means of mono-use needle.
  Arms: 2

SUMMARY:
The incidence of anterior pelvic defect in women is estimated about 10% and it may be often associated to urinary stress incontinence. To date the correction of anterior defects with the use of graft material inserted with transobturator approach has become of large use. Moreover, given the frequent association of urinary stress incontinence to anterior defect, in most of cases it becomes necessary to perform at the same time an anti-incontinence procedure, i.e. a sub-urethral sling positioning. Based on these considerations the aim of this trial will be to compare two different approach for sub-urethral sling positioning, transobturator and transvaginal tape (TOT and TVT) performed in association to transobturator correction of anterior defect with mesh in terms of efficacy and safety.

DETAILED DESCRIPTION:
Women with anterior defect and genuine stress urinary incontinence will be enrolled and randomized in two groups (arm 1 and 2). All patients will be treated with a transobturator correction of anterior defect, in patients of arm 1 will be associated TOT, whereas in patients of arm 2 will be associated TVT.

All patients eligible will undergo baseline assessment consisting of anthropometric, clinical, hormonal, urodynamic, and ultrasonographic evaluations. During the study, the surgical outcomes, the clinical subjective and objective efficacy data, and the adverse experiences will be evaluated in each patient.

Data will be analyzed using the intention-to-treat principle and a P value of 0.05 or less will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Cystocele
* Genuine stress urinary incontinence by self report, examination and test
* Urethral hypermobility
* Eligible for both surgical procedures
* Ambulatory

Exclusion Criteria:

* Pregnancy
* <12 months post-partum
* Systemic disease and/or drugs known to affect bladder function
* Current chemotherapy or radiation therapy
* Urethral diverticulum, augmentation cytoplasty, or artificial sphincter
* Recent pelvic surgery
* Previous pelvic or anti-incontinence surgery
* History of severe abdominopelvic infections
* Known extensive abdominopelvic adhesions
* Detrusor instability and/or intrinsic sphincter dysfunction
* Other gynaecologic pathologies (eg, fibroids, ovarian cysts)
* BMI >30

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-02; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Objective/subjective symptoms improvements | 12 months

SECONDARY OUTCOMES:
Intra-operative complication rate | one day
Postoperative complications rate | 12 months
Failure rate | 12 months
Recurrence rate | 12 months
Quality of life | 12 months
Sexual function | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Palomba, MD, Principal Investigator — Chair of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro; Fulvio Zullo, MD, Study Chair — Chair of Obstetrics and Gynecology, University "Magna Graecia" of Catanzaro
Locations (1):
- "Pugliese" Hospital, Catanzaro, Catanzaro, Italy